CLINICAL TRIAL: NCT06951360
Title: ENERGY Study - Workload Evaluation (Via NASA Task Load Index) of Robotic Assisted and Laparoscopic Surgery
Brief Title: Workload Evaluation (Via NASA Task Load Index) of Robotic Assisted and Laparoscopic Surgery
Acronym: ENERGY
Status: Withdrawn | Type: Observational
Why Stopped: No multicenter recriutiment feasible
Sponsor: Otto-von-Guericke University Magdeburg (Other)
Responsible Party: Principal Investigator, Jessica Stockheim, Dr. med., Otto-von-Guericke University Magdeburg
Other Study IDs: ENERGY study
Record Dates: First submitted 2022-05-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Workplace Stress
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- robotic procedures: residents, specialists and experts performing robotic visceral surgeries
  Interventions: Procedure: ENERGY questionnaire
- laparoscopic procedures: residents, specialists and experts performing laparoscopic visceral surgeries
  Interventions: Procedure: ENERGY questionnaire

INTERVENTIONS:
Procedure: ENERGY questionnaire — Questionnaire including NASA Task Load Index, difficulty level of operation, patient and operation factors

SUMMARY:
workload evaluation (via NASA Task Load Index) of robotic- assisted and laparoscopic surgery

DETAILED DESCRIPTION:
evaluation of individual and overall workload during robotic visceral surgeries using NASA Task Load Index and one additional question referring to difficulty level of the operation in comparison with laparoscopic procedures

ELIGIBILITY:
Inclusion Criteria:

* robotic and laparoscopic procedures

Exclusion Criteria:

* decline of participation (patients, medical stuff)
* paparoscopic appendectomies, laparoscopic cholecystectomies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * involved medical stuff (surgeons, OR nurses, further professions)
  * patients undergoing laparoscopic and robotic procedures fulfilling the inclusion criterias
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Overall workload | 5 years
  NASA Task Load overall workload
surgical expertise | 5 years
  surgical experience counting numbers of open, laparoscopic, robotic procedures and years of surgical practice

SECONDARY OUTCOMES:
NASA Task Load Index subscales | 5 years
  mental, physical, temporal demand, performance, effort, frustration
procedure's difficulty level | 5 years
  additional question to evaluate the variation of difficulty of the performed procedure to expected level of difficulty; 3 levels
patient factors | 5 years
  age, sex, BMI, preexisting illnesses/diseases using CCI (Charlson Comorbidity Index), previous operations, ASA
procedure characteristics | 5 years
  indication, performed operation, intraoperative complications using Clavien-Dindo classification, operation duration, blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Otto-von-Guericke University Magdeburg, Magdeburg, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quan H, Li B, Couris CM, Fushimi K, Graham P, Hider P, Januel JM, Sundararajan V. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. Am J Epidemiol. 2011 Mar 15;173(6):676-82. doi: 10.1093/aje/kwq433. Epub 2011 Feb 17. PMID 21330339
- [Background] Lowndes BR, Forsyth KL, Blocker RC, Dean PG, Truty MJ, Heller SF, Blackmon S, Hallbeck MS, Nelson H. NASA-TLX Assessment of Surgeon Workload Variation Across Specialties. Ann Surg. 2020 Apr;271(4):686-692. doi: 10.1097/SLA.0000000000003058. PMID 30247331